CLINICAL TRIAL: NCT03585348
Title: Importance of Understanding Provider Variability in the Use of Neuromuscular Blocking Drugs and Reversal Agents
Brief Title: Provider Variability in the Use of Neuromuscular Blocking Drugs and Reversal
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Philipp Fassbender, Assistant Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2017P000641; 2017P002631 (Other: Massachusetts General Hospital)
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Neuromuscular Blockade; Residual Curarisation, Postoperative; Surgery Under General Anaesthesia
Keywords: Neuromuscular Blockade Agents; Provider Variability; Quality Improvement; Perioperative Care; Neuromuscular Blockade Reversal
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: The estimated cohort consists of 317.000 adult patients who are intubated for a non-cardiac surgery and extubated at the end of the case at Beth Israel Deaconess Medical Center (205.000) as well as Massachusetts General Hospital (112.000) and received treatment by anesthesia and surgical providers who have completed at least 50 anesthesias and surgeries at their respective institution, respectively.
  Interventions: Other: Neuromuscular blocking agents

INTERVENTIONS:
Other: Neuromuscular blocking agents — Neuromuscular blocking agent ED95 equivalent dose by provider

SUMMARY:
The use of neuromuscular blocking agents during surgery is associated with postoperative respiratory complications and increased risk of readmission to the hospital following ambulatory surgery. Understanding the clinical behavior of providers is essential in devising and assessing quality improvement projects since it is primarily individuals who determine the utilization of neuromuscular blocking drugs and reversal agents, not institutions. Therefore, the primary objective of this study is to determine the variability between individual anesthesia providers (attending physician, resident, nurse anesthetists) in the use of neuromuscular blocking drugs and reversal agents, using advanced statistical methods to adjust for differences in patient and procedure case mix. The investigators hypothesize that variance between individual anesthesia providers in the use of neuromuscular blocking drugs and reversal agents differs depending on provider type.

DETAILED DESCRIPTION:
More than 400 million people receive neuromuscular blocking agents (NMBA) annually, either in the operating theatre to optimize surgical conditions, or in the intensive care unit to facilitate mechanical ventilation in those with patient-ventilator asynchrony. NMBA have been associated with increased morbidity secondary to postoperative residual neuromuscular blockade. The incidence of residual blockade is about 20-60% of patients and depends on compound and dose of NMBA reversal agent used. Despite disagreements over guidelines and thresholds to define the optimal strategy to optimize surgical conditions, there is growing evidence that very high doses of NMBA and neostigmine put the patients at risk of respiratory complications and hospital readmission. The investigators have recently shown that dedicated quality improvement initiatives substantially improve the utilization of non-depolarizing muscle relaxants and their reversal agents.

This is a retrospective, observational, multi-centric cohort study based on on-file hospital data from two institutions, Massachusetts General Hospital and Beth Israel Deaconess Medical Center, Boston, Massachusetts. The investigators will compare the utilization of NMBA cross different groups of anesthesia providers (anesthesiologists, anesthesia residents, CRNAs) who provided anesthesia care in at least 100 cases in their institution. The investigators will control our provider-specific findings for patient-, procedure-, and hospital-specific differences in NMBA utilization.

Primary objective is to determine the variability between individual anesthesia providers in the use of neuromuscular blocking drugs and reversal agents (neostigmine at Massachusetts General Hospital/MGH and neostigmine or sugammadex at Beth Israel Deaconess Medical Center/BIDMC) across provider-types (attending physician, resident, nurse anesthetists (CRNA)), experience level (number of cases done in an institution), and hospitals (MGH, BIDMC).

Potential mechanisms of the provider variability will then be examined, such as providers´age, gender, race, profession, employment status and time of the procedure (surgery conducted during daytime versus nighttime).

Additionally, the investigators will examine if the provider variance in the use of NMBA, neostigmine, and sugammadex (based on mean dose across providers and individual mean dose given for standardized surgical procedures) is associated with respiratory complications and direct costs of care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Non-cardiac surgical procedure
* Endotracheally intubated for surgery and extubated at the end of the case

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Classification Status of 5 or 6
* Other surgery within a month prior to the procedure considered
* Missing covariates

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-cardiac surgical procedure that are intubated for surgery and extubated at the end of the case.
Sampling Method: Non-Probability Sample
Enrollment: 265537 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Neuromuscular blocking agents ED95 equivalent dose or reversal agents dose (neostigmine and/or sugammadex) | During surgery, maximum of 24 hours
  Neuromuscular blocking agent ED95 equivalent dose defined as the median effective dose required to achieve a 95% reduction in maximal twitch response from baseline.

OTHER OUTCOMES:
Respiratory Complications | Up to 7 days after surgery
  Respiratory complications defined as pneumonia, respiratory failure, pulmonary edema, or reintubation.
Direct costs of care | During hospital stay, on average 4 days, and no longer than 1 year
  Direct costs of care defined as costs incurred from admission to discharge day.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Fassbender, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Intercontinental Marketing Services (IMS) Health, Multinational Integrated Data Analysis System (MIDAS), September 2010
- [Background] Thevathasan T, Shih SL, Safavi KC, Berger DL, Burns SM, Grabitz SD, Glidden RS, Zafonte RD, Eikermann M, Schneider JC. Association between intraoperative non-depolarising neuromuscular blocking agent dose and 30-day readmission after abdominal surgery. Br J Anaesth. 2017 Oct 1;119(4):595-605. doi: 10.1093/bja/aex240. PMID 29121289
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Xara D, Silva A, Mendonca J, Abelha F. Inadequate emergence after anesthesia: emergence delirium and hypoactive emergence in the Postanesthesia Care Unit. J Clin Anesth. 2013 Sep;25(6):439-46. doi: 10.1016/j.jclinane.2013.02.011. Epub 2013 Aug 17. PMID 23965209
- [Background] Butterly A, Bittner EA, George E, Sandberg WS, Eikermann M, Schmidt U. Postoperative residual curarization from intermediate-acting neuromuscular blocking agents delays recovery room discharge. Br J Anaesth. 2010 Sep;105(3):304-9. doi: 10.1093/bja/aeq157. Epub 2010 Jun 24. PMID 20576632
- [Background] Lepouse C, Lautner CA, Liu L, Gomis P, Leon A. Emergence delirium in adults in the post-anaesthesia care unit. Br J Anaesth. 2006 Jun;96(6):747-53. doi: 10.1093/bja/ael094. Epub 2006 May 2. PMID 16670111
- [Background] Lien CA, Kopman AF. Current recommendations for monitoring depth of neuromuscular blockade. Curr Opin Anaesthesiol. 2014 Dec;27(6):616-22. doi: 10.1097/ACO.0000000000000132. PMID 25251919
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Brueckmann B, Sasaki N, Grobara P, Li MK, Woo T, de Bie J, Maktabi M, Lee J, Kwo J, Pino R, Sabouri AS, McGovern F, Staehr-Rye AK, Eikermann M. Effects of sugammadex on incidence of postoperative residual neuromuscular blockade: a randomized, controlled study. Br J Anaesth. 2015 Nov;115(5):743-51. doi: 10.1093/bja/aev104. Epub 2015 May 2. PMID 25935840
- [Background] Kotake Y, Ochiai R, Suzuki T, Ogawa S, Takagi S, Ozaki M, Nakatsuka I, Takeda J. Reversal with sugammadex in the absence of monitoring did not preclude residual neuromuscular block. Anesth Analg. 2013 Aug;117(2):345-51. doi: 10.1213/ANE.0b013e3182999672. Epub 2013 Jun 11. PMID 23757472
- [Background] McLean DJ, Diaz-Gil D, Farhan HN, Ladha KS, Kurth T, Eikermann M. Dose-dependent Association between Intermediate-acting Neuromuscular-blocking Agents and Postoperative Respiratory Complications. Anesthesiology. 2015 Jun;122(6):1201-13. doi: 10.1097/ALN.0000000000000674. PMID 25919486
- [Background] Rudolph MI, Chitilian HV, Ng PY, Timm FP, Agarwala AV, Doney AB, Ramachandran SK, Houle TT, Eikermann M. Implementation of a new strategy to improve the peri-operative management of neuromuscular blockade and its effects on postoperative pulmonary complications. Anaesthesia. 2018 Sep;73(9):1067-1078. doi: 10.1111/anae.14326. Epub 2018 Jul 4. PMID 29974459
- [Background] Ladha KS, Bateman BT, Houle TT, De Jong MAC, Vidal Melo MF, Huybrechts KF, Kurth T, Eikermann M. Variability in the Use of Protective Mechanical Ventilation During General Anesthesia. Anesth Analg. 2018 Feb;126(2):503-512. doi: 10.1213/ANE.0000000000002343. PMID 28763357